CLINICAL TRIAL: NCT03761381
Title: Using Optical Coherence Tomography and Noninvasive Retinal Amyloid Imaging to Capture Retinal Changes Associated With Dementia
Brief Title: OCT Angiography and NRAI in Dementia
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, David Huang, MD, PhD, Peterson Professor of Ophthalmology and Professor orf Biomedical Engineering, Oregon Health and Science University
Other Study IDs: IRB#00017045
Record Dates: First submitted 2018-07-02; First posted 2018-12-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease; Dementia; Mild Cognitive Impairment
Keywords: MCI; OCT; Angiography; Alzheimer's; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Early Dementia: This group will consist of adults with suspected dementia/Alzheimer's Disease. OCTA and NRAI data will be gathered in one study visit.
  Interventions: Device: Optical Coherence Tomography Angiography (OCTA) Imaging; Device: Noninvasive Retinal Amyloid Imaging (NRAI)
- Dementia-Free Controls: This group will consist of adults without suspected dementia/Alzheimer's Disease. OCTA and NRAI data will be gathered in one study visit.
  Interventions: Device: Optical Coherence Tomography Angiography (OCTA) Imaging; Device: Noninvasive Retinal Amyloid Imaging (NRAI)

INTERVENTIONS:
Device: Optical Coherence Tomography Angiography (OCTA) Imaging — Optical coherence tomography is a non-invasive imaging technology that provides cross-sectional images of tissues in micron-scale resolution. The angiography component of this device allows for evaluation of blood vessel and blood flow changes in the eye. The Solix device with AngioVue software will be used to detect these blood vessel and flow changes as well as protein deposits in the retinal layers.
Device: Noninvasive Retinal Amyloid Imaging (NRAI) — The Spectralis will be used for NRAI. This system uses a special light source and optical filters to detect fluorescence of amyloid proteins in the eye.

SUMMARY:
The primary goals of this study are to use optical coherence tomography (OCT) angiography (blood vessel mapping) to:

1. Detect retinal blood vessel and blood flow changes in participants with dementia.
2. Detect amyloid protein deposits in the retinas of participants with dementia.

ELIGIBILITY:
Inclusion Criteria for dementia subjects:

* Physician-confirmed diagnosis of probable Alzheimer's disease
* Mild dementia, as defined by score of 20 or greater on the Mini-Mental State Exam, or score of 15 or greater on the Montreal Cognitive Assessment, or Clinical Dementia Rating Scale score of 1.
* Age older than 55 years.
* Able to comply with study procedures
* Corrected visual acuity at least 20/400 in either eye.
* Has a legally authorized representative who can sign study consent form and accompany the participant to the OCT study visit.

Inclusion Criteria for dementia-free controls:

* Age older than 55 years
* Able to comply with study procedures
* Able to maintain stable fixation for OCT imaging
* Corrected visual acuity of at least 20/40 in either eye
* Dementia-free, as defined by score of 24 or greater on the Mini-Mental Status Exam, or a score of 18 or greater on the Montreal Cognitive Assessment, or Clinical Dementia Rating of <1.0.

Exclusion Criteria for both dementia and dementia-free subjects:

* Non-Alzheimer's disease related primary neurologic disease affecting the central nervous system (i.e. multiple sclerosis, Parkinson's disease)
* Evidence on ophthalmological exam within the last year of other ocular diseases or pathology that would confound the assessment of dementia (e.g. glaucoma, diabetic or hypertensive retinal disease, amblyopia, etc.)
* Media opacity such as cataract, corneal scar, or vitreous opacity that could interfere with retinal imaging.
* Previous intraocular surgery except for uncomplicated cataract extraction with posterior chamber intraocular lens implantation
* Inability to maintain stable fixation for OCT imaging or provide informed consent
* Spherical equivalent refractive error greater than +3 or -7 diopters, or astigmatism magnitude of greater than 2 diopters.
* Diabetes for more than 10 years or hemoglobin A1C level of > 10 within the 180 days prior to OCT scanning.
* Uncontrolled hypertension. : SBP > 170 or DBP > 100
* Arrhythmia: irregular pulse, or heart rate not between 50 and 110 beats per minute
* Pregnancy or breast feeding.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dementia subjects will be recruited from the Layton Aging & Alzheimer's Disease Clinic at Oregon Health & Science University. Dementia-free subjects will be recruited from those currently being followed in the Layton Aging & Alzheimer's Disease Center longitudinal aging study with MRI and amyloid PET imaging.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-09-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Retinal amyloid protein detection | 1 day
  OCT and OCT angiography will be used to detect levels of amyloid proteins deposits within the retina layers on the single enrollment visit only. An increase in the protein detection is expected in the dementia group.

SECONDARY OUTCOMES:
Decreased blood flow | 1 day
  OCT and OCT angiography will be used to detect blood flow in dementia vs dementia-free controls. OCT and OCTA imaging will be taken on the single enrollment visit only. Decreased blood flow is expected in the dementia group.
Decreased retinal perfusion | 1 day
  OCT and OCT angiography will be used to detect retinal perfusion deficits in dementia vs dementia-free controls. OCT and OCTA imaging will be taken on a single enrollment visit only. Decreased retinal perfusion is expected in the dementia group.

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States